CLINICAL TRIAL: NCT01521689
Title: Phase II Study of Tolerance and Efficacy of Subcutanous Low Doses Rituximab Given as Consolidation Treatment to Chronic Lymphocytic Leukaemia (CLL) Patients Responding to Induction Therapy
Brief Title: Tolerance and Efficacy of Subcutanous Low Doses Rituximab for CLL Consolidation Treatment
Acronym: LLCRlowdoz
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LLCR lowdoz / IPC 2009-004
Record Dates: First submitted 2011-12-22; First posted 2012-01-31 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: MRD negative CR
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): Consolidation treatment with sub cutaneaous low doses of Rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Low doses of sub cutaneaous rituximab

SUMMARY:
Chronic Lymphocytic Leukemia (CLL) is still an incurable disease. However recent advances have established correlation between the quality of the response (in particular achievement of negativity of minimal residual disease (MRD) and progression free and overall survival. That is why MRD negative complete remission (CR) is the current goal in CLL treatment.

The association of Rituximab fludarabine cyclophosphamide leads to the best response rate with 52 to 72% CR in "medically" fit untreated CLL patients. MRD results in this setting are still preliminary and around 50%. However many other situations (unfit, elderly, relapse, haematological toxicity leading to early interruption of treatment…) are associated with much lower response rate that would be improved by consolidation treatment.

Monoclonal antibodies are the treatment of choice for consolidation because of sparing marrow and targeting CLL cells. Alemtuzumab has been used for this purpose and results confirm improvement of CR and MRD negative responses but alemtuzumab induced immunodeficiency lead to unacceptable infectious complications. Rituximab monotherapy induces low response rate at standard dose regimen. This is at least partially due to shaving of CD20, mechanism by which CD20 is lost from the leukemic cells but these cells are not cleared. Using low doses of rituximab reduced shaving and allowed CLL cells clearance by the mononuclear phagocytic system. Such low doses of rituximab can be administered subcutaneously.

The investigators then propose subcutaneous low dose rituximab in consolidation to CLL patients responding after induction but having not achieved MRD negative CR.

DETAILED DESCRIPTION:
Objective(s) of the clinical study

Main objective:

- To improve the minimal residual disease (MRD) negative complete response (CR) rate after consolidation using subcutaneous low dose of rituximab

Secondary objectives:

* Progression free survival, treatment free survival, overall survival,
* MRD follow-up,
* Safety
* Medico-economic study
* Quality of life study
* Immune functions study (ancillary study)

Main assessment criteria:

MRD negative CR rate, established by peripheral blood 4colour flow cytometry according to international consensus on CLL MRD study, at the end of the consolidation treatment.

Experimental plan:

Inclusion of patients after the evaluation of response to induction treatment according to NCI-ICLLWG criteria and MRD analysis (2 to 3 months after induction completion): patients having not achieved MRD negative CR.

Consolidation treatment by subcutaneous rituximab given at 20 mg/m²/d thrice weekly during 12 weeks.

Evaluation of the response 3 months after completion of the consolidation treatment.

Subjects number: 35 patients will be needed to accept the hypothesis of an augmentation of CR with negative MRD >=40%, excluding the hypothesis that this rate is < 20%. This ensure us an alpha risk at 5% with a 80% power, taking into account that non evaluable patients will be < 5%.

Brief description of the ancillary study:

Immune functions study before and after consolidation treatment by rituximab

ELIGIBILITY:
Inclusion Criteria:

* CLL (Matutes 4 or 5) in CR after induction treatment with negative MRD or PR
* age>18
* performance status<=2
* signed informed consent

Exclusion Criteria:

* cytopenia
* other malignant affection
* HIV or HBV positive
* steroids treatment
* richter syndrome
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Residual disease | up to 3 month after the end of treatment
  - minimal residual disease (MRD) negative complete response (CR) rate after consolidation using subcutaneous low dose of rituximab, from randomisation up to 3 month after the end of treatment

SECONDARY OUTCOMES:
overall survival | From date of inclusion until date of death, assessed up to 10 years
  time between inclusion and death
Adverse events | up to 3 months
  Number and description of adverse events recorded according to the CTC-AE V4
-Quality of life | up to 3 months after the end of treatment
  -Quality of life study by QLQ-C30
Immune functions | up to 3 months after the end of treatment
  NK, monocytes, CD8, and CD 20 expression on leucemic cells or B cells
- Progression free survival | up to time of progression assessed up to 10 years
  Time between inclusion and progression
treatment free survival | up to time of new treatment assessed up to 10 years
  time between end of treatment and restarting a new treatement

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse AURRAN, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

REFERENCES:
- See also: Web site of the sponsor — http://www.institutpaolicalmettes.fr